CLINICAL TRIAL: NCT05160207
Title: Tracheal Intubation-induced Decrease in Heart Rate as an Indicator for Intraoperative Bradycardia During Microlaryngoscopy -a Prospective Observational Trial
Brief Title: Intubation-induced Decrease in Heart Rate as an Indicator for Intraoperative Bradycardia
Status: Completed | Type: Observational
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-10378-BO-ff
Record Dates: First submitted 2021-11-05; First posted 2021-12-16 (Actual); Last update posted 2023-07-19 (Actual); Status verified 2023-07

CONDITIONS: Tracheal Intubation; Airway Management; Heart Rate
Keywords: Laryngoscopy; Bradycardia; Microlaryngoscopy
MeSH Terms: conditions — Bradycardia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This prospective observational study aims to determine, if an tracheal intubation-related decrease in heart rate is associated with intraoperative reflex bradycardia in patients undergoing microlaryngoscopy (MLS) in general anesthesia.

DETAILED DESCRIPTION:
Small studies and case series reported precipitous bradycardia or even asystole due to reflex vagal activity during tracheal intubation and/or laryngoscopy attributable to a so called laryngocardiac reflex (reflex bradycardia); however, larger systematic trials are still lacking. For the purpose of MLS, ENT surgeons frequently apply suspension laryngoscopy (Kleinsasser laryngoscope) in order to visualize the glottis and to enable surgery. Severe bradycardia has been reported during MLS that has been suspected to be induced by reflex vagal activity possibly promoted by the superior laryngeal nerve.

It is still unknown, which patients are at risk for relevant intraoperative bradycardia and moreover, which patients might benefit from preemptive measures such as prophylactic application of positive chronotropic drugs like atropine sulfate, epinephrine or glycopyrrolate. Predictive factors for MLS-induced intraoperative bradycardia have not systematically been investigated yet.

In particularly, it is unknown, if patients that present with a preoperative tracheal intubation-related decrease in heart rate have a predisposition for intraoperative reflex bradycardia during MLS.

This prospective observational study aims to determine, if an tracheal intubation-related decrease in heart rate is associated with intraoperative reflex bradycardia in patients undergoing microlaryngoscopy (MLS) in general anesthesia. Moreover, if we find a positive association, we further aim to determine the predictive value of intubation-relatd bradycardia.

ELIGIBILITY:
Inclusion Criteria:

* Patients requiring general anesthesia with tracheal intubation for elective MLS
* Age ≥ 18

Exclusion Criteria:

* Pregnant or breastfeeding women
* Confirmed indications for awake fiberoptic intubation
* Planned endotracheal intubation without deep anesthesia or neuromuscular blocking agents (e.g. awake videolaryngoscopy)
* Patients at risk for pulmonary aspiration who qualify for rapid sequence induction
* Cardiac pacemaker
* Atrial fibrillation
* Denial of consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients requiring general anesthesia with tracheal intubation for elective MLS in a tertiary care hospital who consent to participate within the study period.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2021-11-04 (Actual); Primary Completion 2022-06-13 (Actual); Study Completion 2022-06-13 (Actual)

PRIMARY OUTCOMES:
Intraoperative decrease of the heart rate | 1 hour
  Continuous intraoperative ECG heart rate measurement (sample rate 1000 hz)

SECONDARY OUTCOMES:
Intraoperative asystolia | 1 hour
  Continuous intraoperative ECG QRS-complex detection (sample rate 1000 hz)
Application of atropine sulfate | 1 hour
  Intraoperative application of atropine sulfate by the responsible anesthetist (yes/no)
Application of positive inotropic drugs | 1 hour
  Intraoperative application of other positive inotropic drugs such as epinephrine by responsible anesthetist (yes/no)
Cardiac arrhythmias | 1 hour
  Continuous intraoperative ECG arrhythmia detection and labeling (sample rate 1000 hz)
Hypotension | 1 hour
  Intraoperative blood pressure measurement
Application of catecholamines or vasoactive drugs | 1 hour
  Intraoperative application of catecholamines or vasoactive drugs by responsible anesthetist (yes/no)
Adverse cardiocirulatory events | 1 hour
  Intraoperative adverse cardiocirulatory events docuimented by the responsible anethetist
PACU stay | 8 hours
  Length of stay in the postanesthesia care unit (PACU)

CONTACTS AND LOCATIONS:
Overall Officials: Martin Petzoldt, MD, Study Chair — Universitätsklinikum Hamburg-Eppendorf; Tanja Peters, Study Chair — Universitätsklinikum Hamburg-Eppendorf; Christian Zöllner, MD, Study Chair — Universitätsklinikum Hamburg-Eppendorf
Locations (1):
- University Medical Center Hamburg-Eppendorf, Hamburg, Germany